CLINICAL TRIAL: NCT03083496
Title: Clinical Evaluation of Different Potassium Oxalate Concentrations in Dentin: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Different Potassium Oxalate Concentrations in Dentin Hypersensitivity Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 61102016.0.0000.5152
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Dentin Sensitivity; Hypersensitivity Dentin; Dentine Hypersensitivity; Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Oxalate 5% (Active Comparator): Prophylaxis of the teeth; an application every 48 hours; 4 sessions
  Interventions: Drug: Potassium Oxalate 5%; Drug: Potassium Oxalate 10%
- Potassium Oxalate 10% (Active Comparator): Prophylaxis of the teeth; an application every 48 hours; 4 sessions
  Interventions: Drug: Potassium Oxalate 5%; Drug: Potassium Oxalate 10%

INTERVENTIONS:
Drug: Potassium Oxalate 5% — Prophylaxis, apply uniformly on the teeth, friccion for 10 seconds, wait 10 minutes, remove the gel from the teeth with cotton and abundant water.
Drug: Potassium Oxalate 10% — Prophylaxis, apply uniformly on the teeth, friccion for 10 seconds, wait 10 minutes, remove the gel from the teeth with cotton and abundant water.

SUMMARY:
This study aims to evaluate the longevity and efficacy of two products potassium oxalate-basedin two concentrations, 10% and 5%, by triple randomized blind clinical trial (split-mouth) . The desensitization approach (single agent) and the long-term effectiveness (baseline, 1 week, 2 weeks, 3 weeks). Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
Dentin hypersensitivity (DH) is characterized as a short, intense and sudden pain caused by thermal, chemical and evaporative stimuli. There are several types of desensitizing agents, used to aid in the control of this pathology, but they are not very effective and have short longevity. The agents based on potassium oxalate have been used by dental surgeons because they have mixed action, both neural and obliterating. Therefore, the aim of this study is through a triple blind randomized clinical trial (split-mouth), evaluate the longevity and efficacy of two products potassium oxalate-based in two concentrations, 10% and 5%. Thirty-two with DH at least 2 teeth and adequate oral hygiene will be randomly divided into two different groups according to the desensitization approach (10% and 5%) The dentin hypersensitivity level will be evaluated immediately after desensitization and after 1, 2 and 3. Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Both genres, interested in the treatment of Dentin Hypersensitivity
* Patients with all teeth in their mouth
* Patients who have at least three teeth with Dentin hypersensitivity in different quadrants
* Good oral hygiene

Exclusion Criteria:

* Caries or unsatisfactory restorations
* Presence of periodontal disease and or parafunctional habits
* Cracks or enamel fractures
* Extensive or unsatisfactory restorations
* Recent restorations involving the labial surface
* Pulpitis
* Dentures
* Orthodontics
* Smokers
* Pregnant women
* Gastroesophageal disease presence
* Uncontrolled systemic disease
* Severe bruxism
* Constant use of analgesic
* Allergic response to dental products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Level of cervical dentin hypersensitivity by using visual analog scale | 3 weeks
  Evaluation of the reduction in dentin hypersensitivity levels by using visual analog scale with a 3 weeks follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo V Soares, DDS,MS,PHD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Paulo V Soares, Uberlândia, Federal University of Uberlandia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grippo JO, Simring M, Coleman TA. Abfraction, abrasion, biocorrosion, and the enigma of noncarious cervical lesions: a 20-year perspective. J Esthet Restor Dent. 2012 Feb;24(1):10-23. doi: 10.1111/j.1708-8240.2011.00487.x. Epub 2011 Nov 17. PMID 22296690
- [Background] Gillam DG, Seo HS, Newman HN, Bulman JS. Comparison of dentine hypersensitivity in selected occidental and oriental populations. J Oral Rehabil. 2001 Jan;28(1):20-5. doi: 10.1046/j.1365-2842.2001.00631.x. PMID 11298905
- [Background] Canadian Advisory Board on Dentin Hypersensitivity. Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. J Can Dent Assoc. 2003 Apr;69(4):221-6. PMID 12662460
- [Background] Brannstrom M. Sensitivity of dentine. Oral Surg Oral Med Oral Pathol. 1966 Apr;21(4):517-26. doi: 10.1016/0030-4220(66)90411-7. No abstract available. PMID 5218158
- [Background] Cunha-Cruz J, Wataha JC, Zhou L, Manning W, Trantow M, Bettendorf MM, Heaton LJ, Berg J. Treating dentin hypersensitivity: therapeutic choices made by dentists of the northwest PRECEDENT network. J Am Dent Assoc. 2010 Sep;141(9):1097-105. doi: 10.14219/jada.archive.2010.0340. PMID 20807910
- [Derived] Galvao ADM, Zeola LF, Moura GF, Teixeira DNR, Gonzaga RCQ, da Silva GR, Soares PV. A long-term evaluation of experimental potassium oxalate concentrations on dentin hypersensitivity reduction: A triple-blind randomized clinical trial. J Dent. 2019 Oct;89:103180. doi: 10.1016/j.jdent.2019.103180. Epub 2019 Aug 12. PMID 31415787